CLINICAL TRIAL: NCT04255810
Title: Systemic Symptoms: Biospecimen Analysis Study
Acronym: BII
Status: Completed | Type: Observational
Sponsor: Glicksman, Caroline, M.D. (Individual)
Collaborators: The Aesthetic Surgery Education & Research Foundation (Other)
Responsible Party: Principal Investigator, Caroline Glicksman, MD and Patricia McGuire, MD, Principle Investigators, The Aesthetic Surgery Education & Research Foundation
Other Study IDs: ASERF-BII Study
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Women With Breast Implants With and Without Self-reported Systemic Symptoms; Women Undergoing an Elective Mastopexy (Breast Lift) or Small Reduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Systemic blood, breast implant capsule tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Women with breast implants and self-reported symptoms of BII: Women undergoing elective breast implant removal without replacement who self-report systemic symptons associated with BII
  Interventions: Procedure: Surgical collection of biospecimens
- Women with breast implants and no self-reported BII: Women undergoing elective breast implant exchange or removal without self-reported symptoms of BII
  Interventions: Procedure: Surgical collection of biospecimens
- Women undergoing elective mastopexy (breast lift): Women undergoing an elective mastopexy (breast lift) without breast implants or soft tissue support

INTERVENTIONS:
Procedure: Surgical collection of biospecimens — Systemic blood and implant capsule tissue will be collected from two cohorts with breast implants, systemic blood only will be collected from Mastopexy cohort
  Groups: Women with breast implants and no self-reported BII; Women with breast implants and self-reported symptoms of BII

SUMMARY:
An increasing number of women are reporting a collection of non-specific systemic symptoms thought to be caused by their breast implants. There is no current pathophysiologic explanation or diagnostic test for BII; it is not a recognized medical disease at this time. This study aims to address the questions asked by patients, physicians, and the FDA with regard to the scientific validity of BII.

DETAILED DESCRIPTION:
An increasing number of women are reporting a collection of non-specific systemic symptoms thought to be caused by their breast implants. The term Breast Implant Illness or "BII" originated with several social media groups. There is no current pathophysiologic explanation or diagnostic test for BII; it is not a recognized medical disease at this time. Recently several studies have been designed and funded to study the role of psychological and social behavioral factors. This study has been designed to scientifically analyze biospecimens from three cohorts of age matched women in the United States. This study aims to address the questions asked by patients, physicians, and the FDA with regard to the scientific validity of BII.

ELIGIBILITY:
Inclusion Criteria:

Consecutive patients who present to investigator surgeon for:

1. Self-reported BII requesting explantation;
2. Patient who presents for breast implant exchange or explantation without self-reported symptoms of BII;
3. Patient who presents for a mastopexy or small reduction less than 200grams (without implants or soft tissue support);
4. Willingness to follow study requirements including 3-6 week and 6 month follow-up exams; and
5. Genetic Female.

Exclusion Criteria:

1. Subject lives more than three hours away from the investigator surgeon;
2. Previous breast reconstruction for cancer;
3. Active malignancy anywhere else in the body;
4. Has been implanted with any silicone implant other than a breast implant anywhere else in the body;
5. History of radiation to the breast;
6. Currently on anti-estrogen therapy; or
7. HIV positive.

Ages: 30 Years to 65 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Genetic females between the ages of 30 and 65 who fall into one of the three cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in self-reported systemic symptoms | 3-6 weeks and 6 months and 1 year
  Change in self-reported symptoms on PROMIS (NIH) questionnaires

CONTACTS AND LOCATIONS:
Locations (1):
- Glicksman Plastic Surgery, Sea Girt, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Anticipated completion of biospecimen and qualitative data collection in 2022, with publication in the Aesthetic Surgery Journal. Four peer reviewed publications in Aesthetic Surgery Journal- ASERF Biospecimen Study.